CLINICAL TRIAL: NCT03161756
Title: A Phase Ib/II Trial of Ipilimumab-Nivolumab-Denosumab and Nivolumab-Denosumab in Patients With Unresectable Stage III and IV Melanoma
Brief Title: Evaluation of Denosumab in Combination With Immune Checkpoint Inhibitors in Patients With Unresectable or Metastatic Melanoma
Acronym: CHARLI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other); Amgen (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01.15
Record Dates: First submitted 2017-05-11; First posted 2017-05-22 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Melanoma Stage Iv; Melanoma Stage Iii; Melanoma
MeSH Terms: conditions — Melanoma | interventions — Denosumab; Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Trial design updated from randomised allocation of patients to physician's choice as per version 2.2 of protocol, there will be a pre-specified number of patients with stage IV M1c disease in each arm (approximately 60%).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental): Patients in Arm A will receive nivolumab 3 mg/kg intravenously (IV) every 2 weeks for 4 doses and denosumab 120 mg subcutaneously (SC) given D1, D8, D15, D29 (induction phase). Thereafter, nivolumab 480 mg IV and denosumab 120 mg SC every 4 weeks for a total of 24 months (maintenance phase).
  Interventions: Drug: Denosumab; Drug: Nivolumab
- Arm B (Experimental): Patients in Arm B will receive ipilimumab at 3 mg/kg combined with nivolumab at 1 mg/kg IV every 3 weeks for 4 doses with denosumab 120 mg SC given D1, D8, D15, D29, D57 (induction phase). This will be followed by nivolumab 480 mg IV and denosumab 120 mg SC ever 4 weeks for a total of 24 months (maintenance phase).
  Interventions: Drug: Denosumab; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Denosumab — Denosumab is a fully human monoclonal immunoglobulin type 2 (IgG2) antibody that binds with high affinity and specificity to RANK ligand (RANKL) and neutralises the activity of human RANKL, similar to the action of endogenous osteoprotegerin (OPG). Denosumab binding prevents the activation of RANK and inhibits the formation, activation, and survival of osteoclasts. As a consequence, bone resorption and cancer-induced bone destruction are reduced.
  Other Names: AMG162
Drug: Nivolumab — Nivolumab is a human monoclonal antibody that targets the programmed death-1 (PD-1) cluster of differentiation 279 (CD279) cell surface membrane receptor. Nivolumab inhibits the interaction of PD-1 with its ligands, PD-L1 and PD-L2, resulting in enhanced T-cell proliferation and interferon-gamma (IFN-γ) release in vitro.
  Other Names: Opdivo; BMS-936558; MDX1106
Drug: Ipilimumab — Ipilimumab is a fully human monoclonal immunoglobulin specific for human cytotoxic T-lymphocyte antigen 4 (CTLA-4), which is expressed on a subset of activated T cells. Ipilimumab is a monoclonal antibody(mAb) that binds to CTLA-4 and blocks the interaction of CTLA-4 with its ligands, cluster of differentiation antigen 80 / cluster of differentiation antigen 86 (CD80 / CD86). Blockade of CTLA-4 has been shown to augment T-cell activation and proliferation, including the activation and proliferation of tumor-infiltrating T-effector cells.
  Other Names: Yervoy; BMS-734016; MDX010
  Arms: Arm B

SUMMARY:
The purpose of this project is to test the addition of a new treatment called denosumab to standard immunotherapies for patients with metastatic melanoma. Denosumab has been used for many years to help treat cancers such as prostate cancer and breast cancer, but it is not currently used in melanoma. We hope the addition of denosumab to current melanoma therapies will make these treatments work better without adding to the side effects.

Who is it for? You may be eligible to join this study if you are aged 18 years or over and have been diagnosed with metastatic melanoma (melanoma that has spread).

Study details: Nivolumab and ipilimumab are approved treatments for advanced melanoma in Australia and overseas. Patients with metastatic melanoma, who are not enrolled in a study, are commonly prescribed nivolumab alone or the combination of nivolumab and ipilimumab as standard care. However, there is limited information on the effectiveness and safety of these treatments in combination with denosumab. Recent melanoma research in animal models has shown that denosumab can make immunotherapies such as ipilimumab and nivolumab work better. Because denosumab has been used in patients with breast and prostate cancer for a long time and is safe, we now want to test the benefits and safety of adding denosumab to immunotherapies in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed unresectable or metastatic melanoma as per AJCC 7 staging system.
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Patient willing and able to provide written informed consent.
5. Treatment naïve (no prior systemic therapy for unresectable or metastatic melanoma). Note that prior adjuvant or neoadjuvant melanoma therapy (except anti-PD1 and/or anti-CTLA-4 therapy) is permitted if it was completed at least 6 weeks prior to allocation, and all related adverse events have either returned to baseline or resolved.
6. Willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.
7. Measurable disease by CT or MRI per RECIST 1.1 criteria.
8. Patients with asymptomatic brain metastasis may be considered for enrollment. These patients can have up to 3 lesions that are ≤ 1.5 cm in diameter. The brain metastasis may be naïve to local therapy or have previously received local therapy (surgery, stereotactic radiotherapy/radiosurgery but not whole brain radiotherapy) and are stable. Asymptomatic from brain metastases at study entry implies that these patients are without corticosteroid, antiepileptics, analgesia or any other treatment for the management of neurological symptoms. Patients with completely resolved neurological symptoms are permitted.
9. At least 2 weeks since the completion of prior therapy, including surgery or radiotherapy.
10. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to registration

    * WBC ≥ 2000/μL
    * Neutrophils ≥ 1500/μL
    * Platelets ≥ 100 x103/μL
    * Haemoglobin > 9.0 g/dL
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

    Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL

    Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
    * AST/ALT ≤ 3 x ULN
    * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
    * Serum calcium of albumin-adjusted calcium ≥ 2.0 mmol/L
11. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug. Appropriate methods of contraception includes:

    * Intrauterine device with a documented failure rate of less than 1% per year.
    * Vasectomised partner who is sterile prior to the female partner patient's commencement of study treatment and is the sole sexual partner for that female.
    * Double barrier contraception: male condom and occlusive cap (diaphragm or cervical /vault caps).
12. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of treatment.
13. Men who are sexually active with a WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with a WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men, do not require contraception. Effective contraception includes:

    * Documented vasectomy and sterility
    * In the partner - intrauterine device with a documented failure rate of less than 1% per year
    * Double barrier contraception: male condom and occlusive cap (diaphragm or cervical/vault caps).
14. Patients must agree to have archival tumour material collected. This can either be from a resected lymph node, primary melanoma, or metastatic site. Where possible, the most recently acquired tumour specimen should be provided. If archival tumour tissue is not available, subjects must consent to allow the acquisition of additional tumour tissue prior to trial entry.
15. Patients enrolled on the biopsy cohort must be agreeable to have serial tumour biopsies during the study.

Exclusion Criteria:

1. Patients are excluded if they have symptomatic, large volume brain metastases and/or any evidence of leptomeningeal disease. Large volume brain metastasis for this study is defined as more than 3 brain metastasis and/or any of the brain metastasis being greater than 1.5 cm in dimension. Note: patients with larger brain metastasis (up to 3 cm) that has been adequately treated with prior surgery or stereotactic radiation are permitted to be enrolled as long as they have adequately recovered from the local therapy.
2. Neurological symptoms from brain metastases present at baseline (resolved neurological symptoms, prior to enrolment, are permitted).
3. Patients with uveal melanoma are excluded.
4. Prior exposure to a CTLA-4 inhibitor (e.g. ipilimumab, tremelimumab), PD-1 inhibitor (e.g. nivolumab, pembrolizumab), PD-L1 inhibitor (e.g. MEDI-4736), PD-L2 inhibitor, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
5. Prior systemic treatment with a BRAF and/or MEK inhibitor
6. Prior treatment with denosumab.
7. Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.
8. Life expectancy of ≤ 6 months.
9. Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw.
10. Active dental or jaw condition, which requires major oral surgery. Patients who have undergone a tooth extraction in less than 4 weeks should be reviewed carefully to ensure they have healed well.
11. Surgery or radiotherapy within less than 2 weeks of Cycle 1 Day 1. Any clinically relevant sequelae from the surgery or radiotherapy must have improved to grade 1 prior to Cycle 1 Day 1.
12. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
13. Patients should be excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enrol if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
14. Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
15. Any investigational drug or other systemic drug therapy for melanoma within 28 days or 5 half-lives from baseline.
16. Pregnant or breastfeeding females.
17. Patients should be excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
18. Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
19. Allergies and Adverse Drug Reaction

    1. History of allergy to study drug components.
    2. History of severe hypersensitivity reaction to any monoclonal antibody.
20. Patients with symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable.
21. For those being registered to Arm B (ipilimumab + nivolumab + denosumab), the use of any vaccines against infectious diseases (e.g. influenza, varicella etc.) within 6 weeks of initiation of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-12-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Median Progression-Free Survival | Approximately 5 years
  Defined as the time from enrolment to date of disease progression as measured using RECIST 1.1 criteria
Occurrence of Grade 3 and 4 Selected Immune-related Adverse Events (irAEs) of interest | Approximately 2 years
  Defined as all irAEs except skin-related toxicity not requiring systemic treatment and laboratory abnormalities not requiring intervention or cessation of treatment with the exception of liver dysfunction and grade 3 thrombocytopenia of greater than 7 days; using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

SECONDARY OUTCOMES:
Rate of Grade 3 and 4 irAEs | Approximately 2 years
  Description of all adverse events by type, frequency and severity using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Best Overall Response According to RECIST 1.1 | Approximately 3 years
  Disease assessment by CT using RECIST v1.1 will be undertaken at Baseline and every 8 weeks (from Week 9) until Week 49 and then every 12 weeks until disease progression.
Progression-Free Survival | Approximately 5 years
  Defined as the time from enrolment to date of disease progression as measured using RECIST 1.1 criteria. Assessed at 6 and 12 months post enrolment.
Overall Survival | Approximately 5 years
  Defined as the time from enrolment to the time of death. Median overall survival will be assessed at 12 and 24 months post enrolment.
Toxicity Profiles of the Checkpoint-Denosumab Combinations | Approximately 2 years
  Description of all adverse events by type, frequency and severity using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Occurrence of Treatment Discontinuation Due to Toxicity | Approximately 2 years
  Number of patients who withdraw from the study due to intolerable adverse reactions

OTHER OUTCOMES:
To assess the local tumour and systemic immunological responses to both combination treatment regimens (exploratory objective) | Approximately 2 years
  As an exploratory objective, this will be done to comprehensively characterise lymphocyte populations residing within the tumour bed and peripheral blood prior to, during and following treatment with RANKL and immune checkpoint inhibition.
To evaluate early FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose) PET (positron emission tomography) response as a predictor of clinical benefit | Approximately 2 years
  As an exploratory objective, this will be done to assess the predictive and prognostic significance of early changes in FDG-PET to immune checkpoint inhibitors and denosumab in conjunction with conventional CT imaging.
To evaluate longitudinal cellular and molecular changes in archival tumour tissue, fresh tumour biopsies and circulating biomarkers to define mechanisms of activity and resistance | Approximately 3 years
  As an exploratory objective, these studies will focus on the mechanism of action of the combination, putative determinants of response and resistance and monitoring of tumour kinetics.
To correlate the makeup and changes in the microbiome with treatment response. | Approximately 2 years
  As an exploratory objective, this is an optional assessment that will allow the collection of samples which will be used to assess and characterise the microbiome in order to better understand determinants of sensitivity and resistance to the study treatments.

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Shahneen Sandhu, Study Chair — Peter MacCallum Cancer Centre, Australia; Prof. Grant McArthur, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (10):
- Australia (10):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Bendigo Health, Bendigo, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No